CLINICAL TRIAL: NCT02418741
Title: The Degree of Neck Flexion Does Not Influence on the Laryngeal View and Discomfort During Endotracheal Intubation in Adult Patients
Brief Title: Head Position for Endotracheal Intubation
Acronym: THHEIEIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Center, Seoul (Other)
Responsible Party: Principal Investigator, Mi Ja Yun, MD, PhD, Principal investigator, National Medical Center, Seoul
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: H-1312/037-002
Record Dates: First submitted 2014-10-12; First posted 2015-04-16 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Intubation; Difficult

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Degree of neck flextion (Experimental): Two degrees of neck flexion were achieved using a 4 cm or 8 cm height of pillow
  Interventions: Other: Neck flexion

INTERVENTIONS:
Other: Neck flexion — Patient's neck was flexed using a 4 cm or 8 cm height of pillow

SUMMARY:
The purpose of this study is to investigate whether degree of neck flexion affect on laryngeal view and discomfort during endotracheal intubation in adult patients.

DETAILED DESCRIPTION:
The neck flexion using a 8 to 10 cm head elevation has been suggested to align laryngeal, pharyngeal and oral axes and facilitate endotracheal intubation by direct laryngoscopy. There have been scarce clinical studies about the appropriate degree of neck flexion for endotracheal intubation. In the present study, the laryngeal view and physician's discomfort during endotracheal intubation were evaluated according to the two degrees of neck flexion(4 cm vs 8 cm) using a 4 or 8 cm height of pillows, respectively, in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Elective operation time ≤2hrs
* American Society of Anesthesiologist, Physical Status 1 or 2
* age ; 18 - 90 years

Exclusion Criteria:

* patient has upper respiratory infection symptoms
* limited mouth opening
* teeth problems
* expecting difficult airway
* congenital heart disease
* patient has a possibility of aspiration pneumonia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Laryngeal view as index of ease of insertion | one year
  Cormack Lehane grade during endotracheal intubation

SECONDARY OUTCOMES:
Discomfort of anesthesiologist during endotracheal intubation | one year
  Anesthesiologist can feel difficulties in mouth opening and in insertion of laryngoscopic blade into oral cavity according to the degrees of neck flexion

CONTACTS AND LOCATIONS:
Overall Officials: Mija Yun, staff, Study Director — National medical center
Locations (1):
- National Medical Center, Seoul, Junggu, South Korea